CLINICAL TRIAL: NCT00640614
Title: Clinical Evaluation of T.R.U.E. TEST® Panel 3.2 Allergens: Gold Sodium Thiosulfate, Hydrocortisone-17-Butyrate, Methyldibromoglutaronitrile, Bacitracin, Parthenolide, Disperse Blue 106, and Bronopol
Brief Title: Clinical Evaluation of T.R.U.E. TEST® : Safety and Efficacy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Allerderm (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Mekos 07 7P3.2 301; 2008-000168-18 (EudraCT Number); WIRB Pr. No.: 20080089 (Other: Western Institutional Review Board)
Record Dates: First submitted 2008-03-03; First posted 2008-03-21 (Estimated); Results first posted 2015-12-22 (Estimated); Last update posted 2020-05-05 (Actual); Status verified 2020-04

CONDITIONS: Contact Dermatitis
Keywords: Dermatitis, Contact
MeSH Terms: conditions — Dermatitis, Contact

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sensitives (Experimental): Subjects with a clinical history and positive patch test (current or previous) to any of the seven allergens. Subjects must otherwise be healthy and fulfill entry criteria.
  Interventions: Biological: T.R.U.E. TEST® Skin Patch Test: Dose Response Allergens
- Consecutives (Experimental): Subjects who are being seen for standard allergy patch testing, that are asked to participate in the study.
  Interventions: Biological: T.R.U.E. TEST® Skin Patch Test: Dose Response Allergens

INTERVENTIONS:
Biological: T.R.U.E. TEST® Skin Patch Test: Dose Response Allergens — Polyvinylpyrrolidone (PVP; excipient 1) Hydrocortisone-17-butyrate, 0.020 mg/cm2 in PVP Hydroxypropylcellulose (HPC; excipient 2) MDBGN, 0.0055 mg/cm2 in PVP Bacitracin, 0.60 mg/cm2 in HPC Gold sodium thiosulfate, 0.075 mg/cm2 in HPC Parthenolide, 0.0030 mg/cm2 in PVP Disperse Blue 106, 0.050 mg/cm2 in PVP Bronopol, 0.25 mg/cm2 in PVP
  Test patches, with allergens, are placed at day one and removed 48 hours later. The duration of the study lasts 21 days. However, the subject is only exposed to the study allergens for 48 hours.
  Other Names: T.R.U.E. TEST® Skin Patch Test: Panel 3.2

SUMMARY:
We propose an open, prospective, multi-center Phase III study to evaluate the diagnostic performance and safety of seven new T.R.U.E. Test allergens: Gold sodium thiosulfate, Hydrocortisone-17-butyrate, Bacitracin, Parthenolide, Methyldibromoglutaronitrile, Disperse blue 106, and Bronopol.Allergen performance and safety will be evaluated in adult patients with suspected contact dermatitis, and in adult patients with a known or suspected sensitization to at least one of the seven allergens.

DETAILED DESCRIPTION:
Primary endpoint:

The performance (efficacy) of each allergen will be evaluated in adult patients with suspected contact dermatitis, and in adult patients with a known or suspected sensitization to at least one of the seven allergens. Performance will be based on:

* Calculated concordance/discordance between T.R.U.E. Test Panel 3.2 allergens and their corresponding petrolatum or aqueous-based allergens.
* Calculated sensitivity and specificity for T.R.U.E. Test Panel 3.2 allergens.

Secondary endpoint:

To evaluate the safety of seven T.R.U.E. Test Panels 3.2 allergens (Gold sodium thiosulfate, Hydrocortisone-17-butyrate, Methyldibromoglutaronitrile, Bacitracin, Parthenolide, Disperse blue 106 and Bronopol) in adult subjects with suspected contact dermatitis ("consecutives"), and/or in adult subjects with a clinical history of contact dermatitis and a current or previous positive patch test to one (or more) of these 7 allergens ("sensitives"). Evaluations will be based on:

* The frequency and characterization of late and/or persistent reactions, tape-induced irritation at the test site, incomplete panel adhesion, and subject-reported sensations of itching or burning during the test period.
* The frequency of adverse events and serious adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Consecutive subjects must report symptoms and/or history consistent with allergic contact dermatitis to at least one of the allergens tested in the study (i.e., subjects are visiting the clinic/physician to diagnose, treat or resolve this condition).
* Sensitive subjects must have a positive patch test to one of the following allergens within the past 10 years.

  * Gold sodium thiosulfate
  * Methyldibromoglutaronitrile (alone or with phenoxyethanol)
  * Bacitracin
  * Bronopol
  * Disperse blue 106 (alone or with Disperse blue 124)
  * Parthenolide (or Compositae mix)
  * Hydrocortisone-17-butyrate
* All subjects must be adults over 18 years of age, and otherwise in good health.
* Premenopausal female subjects with childbearing potential must consent to a urine pregnancy test; urine test results must be negative for study inclusion.
* Informed consent must be signed and understood by each subject, and consistent with all institutional, local and national regulations.

Exclusion Criteria:

* Subjects unable to meet inclusion requirements.
* Women who are breastfeeding or pregnant.
* Topical corticosteroid treatment during the last 7 days before visit 1 on or near the test area.
* Systemic treatment with corticosteroids or other immunosuppressants during the last 7 days.before visit 1.
* Subjects currently receiving (or received in the 21 days before visit 1) other investigational drugs, treatments or devices, or participating in another clinical study.
* Treatment with ultraviolet (UV) light (including tanning) during the 21 days before visit
* Acute dermatitis outbreak or dermatitis on or near the test area on the back.
* Subjects unable to comply with patch test study requirements including multiple return visits and activity restrictions (e.g., protecting test panels from excess moisture due to showering or vigorous activity).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 235 (Actual)
Dates: Start 2008-04; Primary Completion 2009-08 (Actual); Study Completion 2009-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Evy Paulsen, M.D., Ph.D, Principal Investigator — Odense University Hospital; Joseph Fowler, MD, Principal Investigator — Dermatology Specialists PSC; Luz Fonacier, MD, Principal Investigator — Winthrop University; Donald V Belsito, MD, Principal Investigator — American Dermatology Associates; Jerri Hoskyn, MD, Principal Investigator — Rivery City Dermatology; Sandy Skotnicki-Grant, MD, Principal Investigator — Bay Dermatology Centre
Locations (5):
- United States (4):
  - River City Dermatology, Little Rock, Arkansas
  - American Dermatology Associates, Shawnee Mission, Kansas
  - Dermatology Specialists PSC, Louisville, Kentucky
  - Winthrop University Hospital, Mineola, New York
- Odense University Hospital, Odense C, Denmark

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 3 June 2008 through 17 August 2009
Pre-assignment Details: There were no significant events or approaches for the overall study following enrollment but prior to group assignment.
Period: Overall Study
Arm/Group | Sensitives | Consecutives
Started | 125 | 110
Completed | 124 | 110
Not Completed | 1 | 0
Not completed — Lost to Follow-up | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sensitives | Consecutives | Total
Number analyzed (Participants) | 125 | 110 | 235
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 97 | 89 | 186
  >=65 years | 28 | 21 | 49
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.6 (14.93) | 51.2 (14.75) | 50.4 (14.75)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 79 | 78 | 157
  Male | 46 | 32 | 78
Region of Enrollment [Number; unit: participants]
  United States | 97 | 85 | 182
  Canada | 0 | 23 | 23
  Denmark | 28 | 2 | 30

OUTCOME MEASURES:

1. Primary Outcome: Diagnostic Performance: Concordance Between Investigational Allergen and Reference Allergen at Day 21
Description: Concordance: Percentage of subjects who responded positively to T.R.U.E. Test allergen gold sodium thiosulfate and the reference allergen
Time Frame: Visit 5: 21 days after patch application
Population: Subjects with past positive patch test results to gold sodium thiosulfate
Measure: Number (95% Confidence Interval); unit: percentage of concordant responses
Groups:
- Concordance: Percentage of sensitive subjects (per allergen) whose patch test responses were concordant with the reference allergen.
Arm/Group | Concordance
Number analyzed (Participants) | 19
percentage of concordant responses | 78.9 [54.4 to 93.9]

2. Primary Outcome: Diagnostic Performance: Concordance
Description: Concordance: Percentage of subjects who responded positively to T.R.U.E. Test allergen hydrocortisone-17-butyrate and the reference allergen
Time Frame: Visit 5: 21 days after patch application
Population: Subjects with past positive patch test results to hydrocortizone-17-butyrate
Measure: Number (95% Confidence Interval); unit: percentage of concordant responses
Arm/Group | Concordance
Number analyzed (Participants) | 20
percentage of concordant responses | 90 [68.3 to 96.6]

3. Primary Outcome: Diagnostic Performance: Concordance
Description: Concordance: Percentage of subjects who responded positively to T.R.U.E. Test allergen methyldibromo-glutaronitrile and the reference allergen.
Time Frame: Visit 5: 21 days after patch application
Population: Subjects with past positive patch test results to methyldibromo-glutaronitrile
Measure: Number (95% Confidence Interval); unit: percentage of concordant responses
Arm/Group | Concordance
Number analyzed (Participants) | 29
percentage of concordant responses | 62.1 [42.3 to 79.3]

4. Primary Outcome: Diagnostic Performance: Concordance
Description: Concordance: Percentage of subjects who responded positively to TRUE Test allergen bacitracin and the reference allergen.
Time Frame: Visit 5: 21 days after patch application
Population: Subjects with past positive patch test results to bacitracin
Measure: Number (95% Confidence Interval); unit: percentage of concordant responses
Arm/Group | Concordance
Number analyzed (Participants) | 24
percentage of concordant responses | 75 [53.3 to 90.2]

5. Primary Outcome: Diagnostic Performance: Concordance
Description: Concordance: Percentage of subjects who responded positively to TRUE Test allergen parthenolide and the reference allergen.
Time Frame: Visit 5: 21 days after patch application
Population: Subjects with past positive patch test results to parthenolide
Measure: Number (95% Confidence Interval); unit: percentage of concordant responses
Arm/Group | Concordance
Number analyzed (Participants) | 18
percentage of concordant responses | 94.4 [72.7 to 99.9]

6. Primary Outcome: Diagnostic Performance: Concordance
Description: Concordance: Percentage of subjects who responded positively to T.R.U.E. Test allergen disperse blue and the reference allergen.
Time Frame: Visit 5: 21 days after patch application
Population: Subjects with past positive patch test results to disperse blue
Measure: Number (95% Confidence Interval); unit: percentage of concordant responses
Arm/Group | Concordance
Number analyzed (Participants) | 17
percentage of concordant responses | 82.2 [63.6 to 98.5]

7. Primary Outcome: Diagnostic Performance: Concordance
Description: Concordance: Percentage of subjects who responded positively to T.R.U.E. Test allergen bronopol and the reference allergen.
Time Frame: Visit 5: 21 days after patch application
Population: Subjects with past positive test results to bronopol
Measure: Number (95% Confidence Interval); unit: percentage of concordant responses
Arm/Group | Concordance
Number analyzed (Participants) | 23
percentage of concordant responses | 82.6 [61.2 to 95.0]

8. Primary Outcome: Diagnostic Performance: Sensitivity and Specificity: Gold Sodium Thiosulfate
Description: Percentage of subjects with positive (sensitivity) and negative (specificity) results to the investigational allergen and the reference allergen
Time Frame: Visit 5: 21 days after patch application
Measure: Number (95% Confidence Interval); unit: percentage of agreement
Groups:
- Sensitivity: The agreement between positive results for gold sodium thiosulfate and reference allergen
- Specificity: The agreement between the negative results for gold sodium thiosulfate and the reference allergen
Arm/Group | Sensitivity | Specificity
Number analyzed (Participants) | 16 | 16
percentage of agreement | 100 [73.5 to 100] | 57.1 [18.4 to 90.1]

9. Primary Outcome: Diagnostic Performance: Sensitivity and Specificity: Hydrocortisone-17-butyrate
Description: The percentage of subjects with positive (sensitivity) and negative (specificity) results to the investigational allergen and the reference allergen
Time Frame: Visit 5: 21 days after patch application
Measure: Number (95% Confidence Interval); unit: percentage of agreement
Groups:
- Sensitivity: The agreement between positive results for hydrocortisone-17-butyrate and reference allergen
- Specificity: The agreement between negative results for hydrocortisone-17-butyrate and the reference allergen
Arm/Group | Sensitivity | Specificity
Number analyzed (Participants) | 20 | 20
percentage of agreement | 92.3 [64.0 to 99.8] | 85.7 [42.1 to 99.6]

10. Primary Outcome: Diagnostic Performance: Sensitivity and Specificity: Methyldibromo-glutaronitrile
Description: as for outcome 9
Time Frame: Visit 5: 21 days after patch application
Measure: Number (95% Confidence Interval); unit: percentage of agreement
Groups:
- Sensitivity: The agreement between positive results for methyldibromo-glutaronitrile and reference allergen
- Specificity: The agreement between the negative results for methyldibromo-glutaronitrile and the reference allergen
Arm/Group | Sensitivity | Specificity
Number analyzed (Participants) | 29 | 29
percentage of agreement | 28.6 [8.4 to 58.1] | 93.3 [68.1 to 99.8]

11. Primary Outcome: Diagnostic Performance: Sensitivity and Specificity: Bacitracin
Description: as for outcome 9
Time Frame: Visit 5: 21 days after patch application
Measure: Number (95% Confidence Interval); unit: percentage of agreement
Groups:
- Sensitivity: The agreement between positive results for bacitracin and reference allergen
- Specificity: The agreement between the negative results for bacitracin and the reference allergen
Arm/Group | Sensitivity | Specificity
Number analyzed (Participants) | 24 | 24
percentage of agreement | 92.9 [66.1 to 99.8] | 50 [18.7 to 81.3]

12. Primary Outcome: Diagnostic Performance: Sensitivity and Specificity: Parthenolide
Description: as for outcome 9
Time Frame: Visit 5: 21 days after patch application
Measure: Number (95% Confidence Interval); unit: percentage of agreement
Groups:
- Sensitivity: The agreement between positive results for parthenolide and reference allergen
- Specificity: The agreement between negative results for parthenolide and the reference allergen
Arm/Group | Sensitivity | Specificity
Number analyzed (Participants) | 18 | 18
percentage of agreement | 92.9 [66.1 to 99.8] | 100 [39.8 to 100]

13. Primary Outcome: Diagnostic Performance: Sensitivity and Specificity: Disperse Blue
Description: as for outcome 9
Time Frame: Visit 5: 21 days after patch application
Measure: Number (95% Confidence Interval); unit: percentage of agreement
Groups:
- Sensitivity: The agreement between positive results for disperse blue and the reference allergen
- Specificity: The agreement between negative results for disperse blue and the reference allergen
Arm/Group | Sensitivity | Specificity
Number analyzed (Participants) | 15 | 15
percentage of agreement | 88.9 [51.8 to 99.7] | 87.5 [47.3 to 99.7]

14. Primary Outcome: Diagnostic Performance: Sensitivity and Specificity: Bronopol
Description: as for outcome 9
Time Frame: Visit 5: 21 days after patch application
Measure: Number (95% Confidence Interval); unit: percentage of agreement
Groups:
- Sensitivity: The agreement between positive results for bronopol and reference allergen
- Specificity: The agreement between negative results for bronopol and the reference allergen
Arm/Group | Sensitivity | Specificity
Number analyzed (Participants) | 23 | 23
percentage of agreement | 100 [39.8 to 100] | 78.9 [54.4 to 93.9]

15. Secondary Outcome: Safety Evaluations: All T.R.U.E. Test Allergens
Description: Safety Evaluations: Number of participants who experienced Tape Irritation, Itching or Burning and measure of how well patches adhered to the skin.
Time Frame: Day 2: 48 hours after application
Population: NOTE: These secondary measurements apply to the entire subject population and were not separated by 'sensitive' or 'consecutive' subjects.
Measure: Number; unit: participants
Groups:
- Panel Irritation: Irritation from the test panel adhesive and/or tape was scored at day 2 following patch removal
- Itching and Burning: Subject reported sensations of itching and burning were captured at day 2 following patch removal
- Adhesion: Number of subjects whose patches had little to no skin to panel contact prior to removal at visit 2.
Arm/Group | Panel Irritation | Itching and Burning | Adhesion
Number analyzed (Participants) | 235 | 235 | 235
participants | 79 | 123 | 4

16. Secondary Outcome: Late Reactions: All T.R.U.E. Test Allergens
Description: Number of subjects who exhibited Late Reactions (reactions that occur at 7-10 days after application).
Time Frame: 7-10 days after patch application
Measure: Number; unit: participants
Groups:
- Gold Sodium Thiosulfate; Hydrocortisone-17-Butyrate; Methyldibrono-glutaronitrile; Bacitracin; Parthenolide; Disperse Blue; Bronopol: Number of subjects who exhibit reactions 7-10 days after application
Arm/Group | Gold Sodium Thiosulfate | Hydrocortisone-17-Butyrate | Methyldibrono-glutaronitrile | Bacitracin | Parthenolide | Disperse Blue | Bronopol
Number analyzed (Participants) | 234 | 234 | 234 | 234 | 234 | 234 | 234
participants | 6 | 0 | 1 | 0 | 1 | 0 | 0

17. Secondary Outcome: Persistent Reactions: All T.R.U.E. Test Allergens
Description: Number of Subjects who exhibited Persistent Reactions (reactions that initially occur at 2-4 days after application and persist through 7-21 days after application)
Time Frame: initially occur 2-4 days after application and last through 7-21days after patch application
Measure: Number; unit: participants
Arm/Group | Gold Sodium Thiosulfate | Hydrocortisone-17-Butyrate | Methyldibrono-glutaronitrile | Bacitracin | Parthenolide | Disperse Blue | Bronopol
Number analyzed (Participants) | 234 | 234 | 234 | 234 | 234 | 234 | 234
participants | 26 | 6 | 4 | 3 | 12 | 5 | 5

ADVERSE EVENTS:
Time Frame: Day 1 through Day 21
Arm/Group | Sensitives | Consecutives
Serious Adverse Events (participants affected / at risk) | 0/125 | 0/110
Other Adverse Events (participants affected / at risk) | 8/125 | 2/110
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sensitives (N=125) | Consecutives (N=110)
Bruise on mid sternum from motor vehicle accident (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Upper respiratory congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Common head cold symptoms (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Laparoscopic cholecystectomy (Gastrointestinal disorders) | 1 (1) | 0 (0)
Right thumb trauma (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Intense itching (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Intense itching ++ and +++ reactions (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Flare of pre-existing hand eczema during first 3 days of testing (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No